CLINICAL TRIAL: NCT04721379
Title: Impact of Heartfulness Meditation on EEG (Brain Waves) and Meditation Depth
Brief Title: Effect of Heartfulness Meditation on Brain Waves and How Calm One Feels During Meditation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Jay Thimmapuram, Principal Investigator, WellSpan Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1654972
Record Dates: First submitted 2021-01-06; First posted 2021-01-22 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Anxiety; Stress
Keywords: meditation; Heartfulness; EEG; Heart rate
MeSH Terms: conditions — Anxiety Disorders | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into two groups.
  1. Group 1 participants with unguided session simply close their eyes for 10 minutes while EEG and EKG recordings are performed. Following 10 minutes, after briefly opening their eyes, they will be asked to relax with eyes closed for 30 minutes. After finishing the session, they fill out meditation depth questionnaire.
  2. Group 2 participants with guided sessions close their eyes for 10 minutes while EEG and EKG recordings are performed. Following 10 minutes, after briefly opening their eyes, they will be guided through relaxation and meditation session for 30 minutes with a Heartfulness trainer with continued recording. After finishing the session, they also fill out meditation depth questionnaire.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heartfulness Meditation Group (Experimental): Participants will be guided through relaxation and meditation session with a Heartfulness trainer with EEG and EKG recording. After finishing the session, they fill out meditation depth questionnaire.
  Interventions: Behavioral: Meditation
- Control Group with Self Meditation (Active Comparator): Participants will be self-guided through relaxation and meditation session without a trainer with EEG and EKG recording. After finishing the session, they fill out meditation depth questionnaire.
  Interventions: Behavioral: Meditation

INTERVENTIONS:
Behavioral: Meditation — 1. Group 1 participants with unguided session simply close their eyes for 10 minutes while EEG and EKG recordings are performed. Following 10 minutes, after briefly opening their eyes, they will be asked to relax with eyes closed for 30 minutes. After finishing the session, they fill out meditation depth questionnaire.
  2. Group 2 participants with guided sessions close their eyes for 10 minutes while EEG and EKG recordings are performed. Following 10 minutes, after briefly opening their eyes, they will be guided through relaxation and meditation session for 30 minutes with a Heartfulness trainer with continued recording. After finishing the session, they also fill out meditation depth questionnaire.

SUMMARY:
Objectives:

1. To assess the EEG patterns and EKG recordings of participants with no meditation experience with simply closing the eyes for 10 minutes followed by relaxing for 30 minutes.
2. To assess the EEG patterns and EKG recordings of participants with no meditation experience by simply closing the eyes for 10 minutes and then with guided Heartfulness relaxation and meditation for 30 minutes.
3. To assess the baseline anxiety score through GAD-7 questionnaire, subjective experience of all the participants through MEDEQ questionnaire that measures the depth of the meditation experience after the session and correlate with the EEG patterns of the brain and heart rate changes.

EEG and EKG data from the groups will be analyzed by the sleep specialist. EKG device data for HRV and the EEG data will be correlated with the subjective depth of meditation experience in both the groups

DETAILED DESCRIPTION:
Neurological correlates of states of mind during meditation have been studied with Electroencephalogram (EEG) and functional MRIs for many decades. Meditation practices produce distinct EEG brain waveforms, and this may be reflective of the overall subjective experiences. Long term meditators using mindfulness have shown gamma activation on EEG recordings. Practice of Yoganidra and Sahaja meditation have been reported to show increased theta activity. Transcendental Meditation practices have shown alpha waves during meditative periods. While most of the meditative practices may appear similar, there may be subtle differences that might make them better suited for particular conditions. However, most of the studies conducted were small, non-randomized and therefore the outcomes are unclear.

The investigators wish to conduct a randomized controlled prospective study using Heartfulness meditation techniques. Heartfulness meditation practice is a simple heart-based meditation practice that has been shown to improve burnout, emotional wellness and sleep. In a younger subset of patients, it has also shown to increase the telomere length. However, the neurological and physiological correlates of this practice have not been assessed. This study will investigate whether using this novel approach of a heart-based meditation program leads to measurable changes in the EEG and also whether there is any correlation with the waveforms and the depth of meditation. This may provide an explanation from a neurological basis for the improvement of certain wellness parameters such as sleep. In addition, meditation practices have been shown to have positive benefits on cardiovascular system including heart rate variability (HRV). Cardiovascular physiology measured by continuous electrocardiogram (EKG) monitoring is a non-invasive way of measuring HRV. In this study, a correlation of the EEG and HRV with the subjective depth of meditation experience measured through meditation depth questionnaire (MEDEQ) along with baseline anxiety score as measured by generalized anxiety disorder scale (GAD-7) will be assessed.

Primary outcome and Hypotheses:

1. The primary outcome will be observing a change in EEG pattern of subjects who follow a Heartfulness guided meditation as compared to unguided self-relaxation and meditation.
2. The study team hypothesize that guided Heartfulness meditation will be associated with deeper relaxed brain wave patterns - predominantly theta and delta waves - compared to beta and alpha waves in unguided self-relaxation and meditation. The investigators anticipate that subjects will perceive an increased depth of meditation during a guided relaxation session compared to simply closing the eyes for the duration of the study. Since participants have no prior meditation experience, the investigators hypothesize that the first attempt at meditation is adequate to induce a relaxed state and EEG changes.
3. With regards to EKG changes, the study team hypothesize that there will be a reduction in heart rate and increased beat-to-beat variability with guided meditation as compared to unguided self-relaxation for the same duration.

ELIGIBILITY:
Inclusion Criteria:

• Adults above 18 years of age willing to participate in the study.

Exclusion Criteria:

* Participants unwilling to participate in the study and those with prior meditation experience.
* Participants who are unable to sit for 30 minutes due to either physical or mental conditions will be excluded.
* Participants with bipolar disorder, substance abuse (drugs or alcohol abuse in last 6 months), alcohol withdrawal, BMI < 18, suicidal ideation, active psychotherapy, major depression, anxiety disorder, obstructive sleep apnea, eating disorder, history of brain surgery or known brain tumors, known seizures or on treatment for seizures, borderline personality disorder, post-traumatic stress disorder, or psychotic disorder.
* Participants with known heart rhythm problems such as atrial fibrillation is advised not to participate.
* Participants on benzodiazepines or psychiatry medications, stimulants or sleeping pills that may potentially interfere with EEG patterns will be excluded.
* Participants on cardiovascular medications that affect the heart rate will be excluded.
* Participants who are unable to have the leads on their scalp or skin will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2022-08-15 (Estimated); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Brain wave changes with Heartfulness guided meditation comparing with self-guided meditation | Through completion of study, average of one hour.
  During meditation, EEG will be recorded using brain wave leads.
EKG changes with Heartfulness guided meditation comparing with self-guided meditation | Through completion of study, average of one hour.
  During meditation, EKG will be recorded using chest leads.
Meditation depth Index questionnaire with Heartfulness guided meditation comparing with self-guided meditation | After the meditation session, average of 10 minutes
  The questionnaire will be completed after the 10 minute meditation session and again after 30 minute meditation session

SECONDARY OUTCOMES:
Generalized Anxiety score | Before the meditation session, average of 5 minutes.
  Using Generalized Anxiety Disorder -7 score. Scores 5-9 indicate mild anxiety, 10-14 indicate moderate anxiety and 15-21 indicate severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- WellSpan Dover Sleep Center, Dover, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No